CLINICAL TRIAL: NCT02285595
Title: A Prospective, Multicenter Study Comparing Healing After Treatment With the Sonendo GentleWave™ System as Compared to a Traditional Root Canal Therapy Literature Control
Brief Title: Sonendo GentleWave™ System for Treatment in Molar Teeth Requiring Root Canal Therapy
Acronym: SUPREME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonendo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-06
Record Dates: First submitted 2014-11-03; First posted 2014-11-07 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Root Canal Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (1):
- Sonendo GentleWave™ System (Other): The Sonendo GentleWave System is intended to prepare, clean, and irrigate 1st and 2nd molar teeth indicated for root canal therapy.
  Interventions: Device: Sonendo GentleWave™ System

INTERVENTIONS:
Device: Sonendo GentleWave™ System

SUMMARY:
A prospective, literature controlled, clinical study evaluating healing rates for the Sonendo GentleWave System in the treatment of 1st and 2nd molars indicated for root canal therapy.

DETAILED DESCRIPTION:
A prospective, non-significant risk device, literature controlled, study evaluating healing rates for the Sonendo GentleWave System in the treatment of 1st and 2nd molars indicated for root canal therapy.

All patients will receive root canal therapy with the Sonendo GentleWave System. All patients will be followed for 24 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Indicated for root canal therapy
* First or second molar
* Signed informed consent form

Exclusion Criteria:

* Poor oral hygiene
* Class II or III mobility
* Open or incompletely formed root apices
* Vertical fracture, horizontal fracture, or perforation below the Cemento-Enamel Junction (CEJ)
* Previous pulpectomy or root canal therapy

Note: Additional exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Miller, Study Director — Sonendo, Inc.
Locations (3):
- United States (3):
  - Shahriar Rassoulian, DMD, Aliso Viejo, California
  - Khang Le, DDS, Santa Ana, California
  - Stacey Woo, DDS, Whittier, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters OA, Schonenberger K, Laib A. Effects of four Ni-Ti preparation techniques on root canal geometry assessed by micro computed tomography. Int Endod J. 2001 Apr;34(3):221-30. doi: 10.1046/j.1365-2591.2001.00373.x. PMID 12193268
- [Background] Peters OA, Peters CI, Schonenberger K, Barbakow F. ProTaper rotary root canal preparation: effects of canal anatomy on final shape analysed by micro CT. Int Endod J. 2003 Feb;36(2):86-92. doi: 10.1046/j.1365-2591.2003.00626.x. PMID 12657151
- [Background] Shuping GB, Orstavik D, Sigurdsson A, Trope M. Reduction of intracanal bacteria using nickel-titanium rotary instrumentation and various medications. J Endod. 2000 Dec;26(12):751-5. doi: 10.1097/00004770-200012000-00022. PMID 11471648
- [Background] McGurkin-Smith R, Trope M, Caplan D, Sigurdsson A. Reduction of intracanal bacteria using GT rotary instrumentation, 5.25% NaOCl, EDTA, and Ca(OH)2. J Endod. 2005 May;31(5):359-63. doi: 10.1097/01.don.0000145035.85272.7c. PMID 15851929
- [Background] Hulsmann M, Schade M, Schafers F. A comparative study of root canal preparation with HERO 642 and Quantec SC rotary Ni-Ti instruments. Int Endod J. 2001 Oct;34(7):538-46. doi: 10.1046/j.1365-2591.2001.00431.x. PMID 11601772
- [Background] Vaudt J, Bitter K, Neumann K, Kielbassa AM. Ex vivo study on root canal instrumentation of two rotary nickel-titanium systems in comparison to stainless steel hand instruments. Int Endod J. 2009 Jan;42(1):22-33. doi: 10.1111/j.1365-2591.2008.01489.x. PMID 19125977
- [Background] Wilcox LR, Roskelley C, Sutton T. The relationship of root canal enlargement to finger-spreader induced vertical root fracture. J Endod. 1997 Aug;23(8):533-4. doi: 10.1016/S0099-2399(97)80316-0. PMID 9587326
- [Background] Wu MK, R'oris A, Barkis D, Wesselink PR. Prevalence and extent of long oval canals in the apical third. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Jun;89(6):739-43. doi: 10.1067/moe.2000.106344. PMID 10846130
- [Background] Jafarzadeh H, Abbott PV. Ledge formation: review of a great challenge in endodontics. J Endod. 2007 Oct;33(10):1155-62. doi: 10.1016/j.joen.2007.07.015. Epub 2007 Sep 4. PMID 17889681
- [Background] Cohen S., Burns R. C. Pathways of the pulp. 8th ed. St Louis: Mosby, 2002.
- [Background] Kapalas A, Lambrianidis T. Factors associated with root canal ledging during instrumentation. Endod Dent Traumatol. 2000 Oct;16(5):229-31. doi: 10.1034/j.1600-9657.2000.016005229.x. PMID 11202887
- [Background] Harty FJ, Parkins BJ, Wengraf AM. Success rate in root canal therapy. A retrospective study of conventional cases. Br Dent J. 1970 Jan 20;128(2):65-70. doi: 10.1038/sj.bdj.4802429. No abstract available. PMID 5270224
- [Background] Namazikhah MS, Mokhlis HR, Alasmakh K. Comparison between a hand stainless-steel K file and a rotary NiTi 0.04 taper. J Calif Dent Assoc. 2000 Jun;28(6):421-6. PMID 11324127
- [Background] Greene KJ, Krell KV. Clinical factors associated with ledged canals in maxillary and mandibular molars. Oral Surg Oral Med Oral Pathol. 1990 Oct;70(4):490-7. doi: 10.1016/0030-4220(90)90217-g. PMID 2216387
- [Background] Gutmann J. L., Dumsha T. C., Lovdahl P. E., Hovland E. J. Problem Solving in Endodontics (3rd ed.). St. Louis: Mosby, 1997.
- [Background] Bergenholtz G, Lekholm U, Milthon R, Heden G, Odesjo B, Engstrom B. Retreatment of endodontic fillings. Scand J Dent Res. 1979 Jun;87(3):217-24. doi: 10.1111/j.1600-0722.1979.tb00675.x. PMID 293884
- [Background] Stadler LE, Wennberg A, Olgart L. Instrumentation of the curved root canal using filing or reaming technique--a clinical study of technical complications. Swed Dent J. 1986;10(1-2):37-43. PMID 3458317
- [Background] Eleftheriadis GI, Lambrianidis TP. Technical quality of root canal treatment and detection of iatrogenic errors in an undergraduate dental clinic. Int Endod J. 2005 Oct;38(10):725-34. doi: 10.1111/j.1365-2591.2005.01008.x. PMID 16164687
- [Background] Seltzer S, Bender IB, Smith J, Freedman I, Nazimov H. Endodontic failures--an analysis based on clinical, roentgenographic, and histologic findings. I. Oral Surg Oral Med Oral Pathol. 1967 Apr;23(4):500-16. doi: 10.1016/0030-4220(67)90546-4. No abstract available. PMID 5227403
- [Background] Alhadainy HA. Root perforations. A review of literature. Oral Surg Oral Med Oral Pathol. 1994 Sep;78(3):368-74. doi: 10.1016/0030-4220(94)90070-1. PMID 7970600
- [Background] Jew RC, Weine FS, Keene JJ Jr, Smulson MH. A histologic evaluation of periodontal tissues adjacent to root perforations filled with Cavit. Oral Surg Oral Med Oral Pathol. 1982 Jul;54(1):124-35. doi: 10.1016/0030-4220(82)90427-3. PMID 6956820
- [Background] Ingle J. I., Bakland L. K. Endodontics. 5th ed. London: BC Decker Inc., 2002.
- [Background] Swartz DB, Skidmore AE, Griffin JA Jr. Twenty years of endodontic success and failure. J Endod. 1983 May;9(5):198-202. doi: 10.1016/S0099-2399(83)80092-2. No abstract available. PMID 6574207
- [Background] Sjogren U, Hagglund B, Sundqvist G, Wing K. Factors affecting the long-term results of endodontic treatment. J Endod. 1990 Oct;16(10):498-504. doi: 10.1016/S0099-2399(07)80180-4. PMID 2084204
- [Background] Smith CS, Setchell DJ, Harty FJ. Factors influencing the success of conventional root canal therapy--a five-year retrospective study. Int Endod J. 1993 Nov;26(6):321-33. doi: 10.1111/j.1365-2591.1993.tb00765.x. PMID 8144241
- [Background] Friedman S, Lost C, Zarrabian M, Trope M. Evaluation of success and failure after endodontic therapy using a glass ionomer cement sealer. J Endod. 1995 Jul;21(7):384-90. doi: 10.1016/S0099-2399(06)80976-3. PMID 7499981
- [Background] ElAyouti A, Weiger R, Lost C. Frequency of overinstrumentation with an acceptable radiographic working length. J Endod. 2001 Jan;27(1):49-52. doi: 10.1097/00004770-200101000-00018. PMID 11487165
- [Background] ElAyouti A, Dima E, Ohmer J, Sperl K, von Ohle C, Lost C. Consistency of apex locator function: a clinical study. J Endod. 2009 Feb;35(2):179-81. doi: 10.1016/j.joen.2008.10.017. Epub 2008 Dec 12. PMID 19166768
- [Background] Williams CB, Joyce AP, Roberts S. A comparison between in vivo radiographic working length determination and measurement after extraction. J Endod. 2006 Jul;32(7):624-7. doi: 10.1016/j.joen.2005.10.044. PMID 16793467
- [Background] Parashos P, Gordon I, Messer HH. Factors influencing defects of rotary nickel-titanium endodontic instruments after clinical use. J Endod. 2004 Oct;30(10):722-5. doi: 10.1097/01.don.0000129963.42882.c9. PMID 15448468
- [Background] Parashos P, Messer HH. Rotary NiTi instrument fracture and its consequences. J Endod. 2006 Nov;32(11):1031-43. doi: 10.1016/j.joen.2006.06.008. PMID 17055902
- [Background] Suter B, Lussi A, Sequeira P. Probability of removing fractured instruments from root canals. Int Endod J. 2005 Feb;38(2):112-23. doi: 10.1111/j.1365-2591.2004.00916.x. PMID 15667633
- [Background] Seltzer S, Naidorf IJ. Flare-ups in endodontics: I. Etiological factors. J Endod. 1985 Nov;11(11):472-8. doi: 10.1016/S0099-2399(85)80220-X. No abstract available. PMID 3868692
- [Background] Naidorf IJ. Endodontic flare-ups: bacteriological and immunological mechanisms. J Endod. 1985 Nov;11(11):462-4. doi: 10.1016/S0099-2399(85)80218-1. No abstract available. PMID 3868690
- [Background] Vande Visse JE, Brilliant JD. Effect of irrigation on the production of extruded material at the root apex during instrumentation. J Endod. 1975 Jul;1(7):243-6. doi: 10.1016/s0099-2399(75)80227-5. No abstract available. PMID 1061800
- [Background] Martin H, Cunningham WT. The effect of endosonic and hand manipulation on the amount of root canal material extruded. Oral Surg Oral Med Oral Pathol. 1982 Jun;53(6):611-3. doi: 10.1016/0030-4220(82)90350-4. No abstract available. PMID 6954443
- [Background] al-Omari MA, Dummer PM. Canal blockage and debris extrusion with eight preparation techniques. J Endod. 1995 Mar;21(3):154-8. doi: 10.1016/s0099-2399(06)80443-7. PMID 7561660
- [Background] Reddy SA, Hicks ML. Apical extrusion of debris using two hand and two rotary instrumentation techniques. J Endod. 1998 Mar;24(3):180-3. doi: 10.1016/S0099-2399(98)80179-9. PMID 9558583
- [Background] Ferraz CC, Gomes NV, Gomes BP, Zaia AA, Teixeira FB, Souza-Filho FJ. Apical extrusion of debris and irrigants using two hand and three engine-driven instrumentation techniques. Int Endod J. 2001 Jul;34(5):354-8. doi: 10.1046/j.1365-2591.2001.00394.x. PMID 11482718
- [Background] Azar NG, Ebrahimi G. Apically-extruded debris using the ProTaper system. Aust Endod J. 2005 Apr;31(1):21-3. doi: 10.1111/j.1747-4477.2005.tb00202.x. PMID 15881729
- [Background] Tinaz AC, Alacam T, Uzun O, Maden M, Kayaoglu G. The effect of disruption of apical constriction on periapical extrusion. J Endod. 2005 Jul;31(7):533-5. doi: 10.1097/01.don.0000152294.35507.35. PMID 15980716
- [Background] Tanalp J, Kaptan F, Sert S, Kayahan B, Bayirl G. Quantitative evaluation of the amount of apically extruded debris using 3 different rotary instrumentation systems. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Feb;101(2):250-7. doi: 10.1016/j.tripleo.2005.03.002. Epub 2005 Oct 14. PMID 16448929
- [Background] Kustarci A, Akpinar KE, Er K. Apical extrusion of intracanal debris and irrigant following use of various instrumentation techniques. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Feb;105(2):257-62. doi: 10.1016/j.tripleo.2007.06.028. PMID 18230395
- [Background] Logani A, Shah N. Apically extruded debris with three contemporary Ni-Ti instrumentation systems: an ex vivo comparative study. Indian J Dent Res. 2008 Jul-Sep;19(3):182-5. doi: 10.4103/0970-9290.42947. PMID 18797091
- [Background] Salzgeber RM, Brilliant JD. An in vivo evaluation of the penetration of an irrigating solution in root canals. J Endod. 1977 Oct;3(10):394-8. doi: 10.1016/S0099-2399(77)80172-6. No abstract available. PMID 270543
- [Background] Balto H., Al-Nazhan S. s.l, Accidental injection of sodium hypochlorite beyond the root apex: Saudi Dent. J., 2002, Vol. 14.
- [Background] Becker GL, Cohen S, Borer R. The sequelae of accidentally injecting sodium hypochlorite beyond the root apex. Report of a case. Oral Surg Oral Med Oral Pathol. 1974 Oct;38(4):633-8. doi: 10.1016/0030-4220(74)90097-8. No abstract available. PMID 4547330
- [Background] Becking AG. Complications in the use of sodium hypochlorite during endodontic treatment. Report of three cases. Oral Surg Oral Med Oral Pathol. 1991 Mar;71(3):346-8. doi: 10.1016/0030-4220(91)90313-2. PMID 2011360
- [Background] Bowden JR, Ethunandan M, Brennan PA. Life-threatening airway obstruction secondary to hypochlorite extrusion during root canal treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):402-4. doi: 10.1016/j.tripleo.2005.06.021. Epub 2005 Oct 5. No abstract available. PMID 16504876
- [Background] Cymbler DM, Ardakani P. Sodium hypochlorite injection into periapical tissues. Dent Update. 1994 Oct;21(8):345-6. PMID 7641958
- [Background] Ehrich DG, Brian JD Jr, Walker WA. Sodium hypochlorite accident: inadvertent injection into the maxillary sinus. J Endod. 1993 Apr;19(4):180-2. doi: 10.1016/S0099-2399(06)80684-9. PMID 8326264
- [Background] Gatot A, Arbelle J, Leiberman A, Yanai-Inbar I. Effects of sodium hypochlorite on soft tissues after its inadvertent injection beyond the root apex. J Endod. 1991 Nov;17(11):573-4. doi: 10.1016/S0099-2399(06)81725-5. PMID 1812208
- [Background] Herrmann JW, Heicht RC. Complications in therapeutic use of sodium hypochlorite. J Endod. 1979 May;5(5):160. doi: 10.1016/S0099-2399(79)80039-4. No abstract available. PMID 296258
- [Background] Hulsmann M, Hahn W. Complications during root canal irrigation--literature review and case reports. Int Endod J. 2000 May;33(3):186-93. doi: 10.1046/j.1365-2591.2000.00303.x. PMID 11307434
- [Background] Joffe E. Complication during root canal therapy following accidental extrusion of sodium hypochlorite through the apical foramen. Gen Dent. 1991 Nov-Dec;39(6):460-1. No abstract available. PMID 1813356
- [Background] Kavanagh CP, Taylor J. Inadvertent injection of sodium hypochlorite into the maxillary sinus. Br Dent J. 1998 Oct 10;185(7):336-7. doi: 10.1038/sj.bdj.4809809. PMID 9807916
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Gracely RH, Kwilosz DM. The Descriptor Differential Scale: applying psychophysical principles to clinical pain assessment. Pain. 1988 Dec;35(3):279-288. doi: 10.1016/0304-3959(88)90138-8. PMID 3226757
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Background] Louis H. Berman and Gary R. Hartwell. "Diagnosis", in pathways of the Pulp, K. Hargreaves, S. Cohen, 10th ed. St. Louis: Mosby, 2011.
- [Background] Berman L. H., Hartwell, G. R. "Diagnosis", in Pathways of the Pulp, ed. S. Cohen, K. Hargreaves, 9th ed. St. Louis: Mosby, 2006.
- [Background] Harpenau, L. A. "Furcation Involvement", in Hall's Critical Decisions in Periodontology, ed. Harpenau, L. A. Shelton, CT: People's Medical Publishing House, 2013.
- [Background] Glickman GN. AAE Consensus Conference on Diagnostic Terminology: background and perspectives. J Endod. 2009 Dec;35(12):1619-20. doi: 10.1016/j.joen.2009.09.029. No abstract available. PMID 19932336
- [Background] Tani-Ishii N, Teranaka T. Clinical and radiographic evaluation of root-canal obturation with obtura II. J Endod. 2003 Nov;29(11):739-42. doi: 10.1097/00004770-200311000-00013. PMID 14651281
- [Background] de Sermeno RF, da Silva LA, Herrera H, Herrera H, Silva RA, Leonardo MR. Tissue damage after sodium hypochlorite extrusion during root canal treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Jul;108(1):e46-9. doi: 10.1016/j.tripleo.2008.12.024. Epub 2009 May 13. PMID 19442541
- [Background] Koseoglu BG, Tanrikulu S, Subay RK, Sencer S. Anesthesia following overfilling of a root canal sealer into the mandibular canal: a case report. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Jun;101(6):803-6. doi: 10.1016/j.tripleo.2005.07.015. Epub 2006 Jan 4. PMID 16731404
- [Background] Sari S, Duruturk L. Radiographic evaluation of periapical healing of permanent teeth with periapical lesions after extrusion of AH Plus sealer. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Sep;104(3):e54-9. doi: 10.1016/j.tripleo.2007.03.024. PMID 17709070
- [Background] World Medical Association.. World Medical Association Declaration of Helsinki. Ethical principles for medical research involving human subjects. Bull World Health Organ. 2001;79(4):373-4. Epub 2003 Jul 2. No abstract available. PMID 11357217

RESULTS

PARTICIPANT FLOW:
Groups:
- GentleWave™ Treatment Group: Participants were given Sonendo GentleWave System Root Canal Treatment to prepare, clean, and irrigate 1st and 2nd molar teeth indicated for root canal therapy.
Period: Overall Study
Arm/Group | GentleWave™ Treatment Group
Started | 69
Completed | 54
Not Completed | 15
Not completed — Lost to Follow-up | 14
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GentleWave™ Treatment Group
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race of Participants: Asian | 8
  Race of Participants: Black/ African American | 3
  Race of Participants: Caucasian | 20
  Race of Participants: Hispanic | 36
  Race of Participants: Other | 2
PAI Score [Count of Participants; unit: Participants] — Orstavik D., Kerekes K, Ericksen H. M. The periapical index: A scoring system for radiographic assessment of apical periodontitis. Dent Traumatol J 1986;2: 20-34.
  Score of 1: Normal Score of 2: Small changes in bone structure Score of 3: Changes in bone structure with some mineral loss (bone loss) Score of 4: Periodontitis with well-defined radiolucent area (apical periodontitis) Score of 5: Severe Periodontitis with exacerbating features (apical periodontitis) Population: One subject had withdrawn from the study prior to data analysis. Healed is defined by absence of a radiographic indication of apical peridontitis (PAI <3) and absence of clinical signs and symptoms other than tenderness to percussion.
  Participants
    number analyzed (Participants) | 68
    PAI Score < 3 | 43
    PAI Score = 3 | 16
    PAI Score 4 or 5 | 9
Periradicular Diagnosis [Count of Participants; unit: Participants] — AAE Consensus Conference Recommended Diagnostic Terminology, JOE 35(12):1634, 2009.
  Symptomatic Apical Periodontitis: Inflammation, with clinical symptoms. Asymptomatic Apical Periodontitis: Inflammation with apical radiolucent area, does not produce clinical symptoms.
  Acute Apical Abscess: Inflammation characterized by rapid onset of clinical symptoms and swelling.
  Chronic Apical Abscess: Inflammation characterized by gradual onset, little or no discomfort, presence of a sinus tract.
  Condensing Osteitis: Diffuse radiopaque lesion representing a localized bony reaction to inflammation. Population: One patient withdrew prior to data analysis
  Participants
    number analyzed (Participants) | 68
    Normal periradicular tissue | 12
    Healing within normal limits | 0
    Symptomatic apical periodontitis | 39
    Asymptomatic apical periodontitis | 11
    Acute Apical Abscess | 2
    Chronic Apical Abscess | 3
    Condensing Osteitis | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a PAI Score of < 3, = 3, or = 4 or 5
Description: The periapical index: A scoring system for radiographic assessment of apical periodontitis. Score of 1: Normal. Score of 2: Small changes in bone structure. Score of 3: Changes in bone structure with some mineral loss (bone loss). Score of 4: Periodontitis with well-defined radiolucent area (apical periodontitis). Score of 5: Severe Periodontitis with exacerbating features (apical periodontitis).
  Healed is defined by absence of a radiographic indication of apical periodontitis (PAI <3) and absence of clinical signs and symptoms other than tenderness to percussion.
  Healing is defined by a reduction of radiolucency (if radiolucency is present at Baseline) combined with the absence of clinical signs and symptoms other than tenderness to percussion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | GentleWave™ Treatment Group
Number analyzed (Participants) | 54
Participants
  PAI Score < 3 | 51
  PAI Score = 3 | 3
  PAI Score 4 or 5 | 0

2. Primary Outcome: Periradicular Diagnosis
Description: Symptomatic Apical Periodontitis: Inflammation, with clinical symptoms. Asymptomatic Apical Periodontitis: Inflammation with apical radiolucent area, does not produce clinical symptoms. Acute Apical Abscess: Inflammation characterized by rapid onset of clinical symptoms and swelling. Chronic Apical Abscess: Inflammation characterized by gradual onset, little or no discomfort, presence of a sinus tract. Condensing Osteitis: Diffuse radiopaque lesion representing a localized bony reaction to inflammation. Healed is defined by absence of a radiographic indication of apical periodontitis (PAI <3) and absence of clinical signs and symptoms other than tenderness to percussion.
  Healing is defined by a reduction of radiolucency (if radiolucency is present at Baseline) combined with the absence of clinical signs and symptoms other than tenderness to percussion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | GentleWave™ Treatment Group
Number analyzed (Participants) | 54
Participants
  Normal Apical Tissue | 40
  Symptomatic Apical Periodontitis | 0
  Asymptomatic Apical Periodontitis | 0
  Acute Apical Abscess | 0
  Chronic Apical Abscess | 0
  Condensing Osteitis | 0
  Healing Within Normal Limits | 14

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | GentleWave™ Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT02285595/Prot_SAP_000.pdf